CLINICAL TRIAL: NCT04279496
Title: Coronary CT Angiography Evaluation for Clinical Outcomes: An International Multicenter
Brief Title: Coronary CT Angiography Evaluation for Clinical Outcomes: An International Multicenter Registry
Acronym: CONFIRM2
Status: Enrolling by invitation | Type: Observational
Sponsor: Cleerly, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Confirm2-Registry
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective of CONFIRM2 is to perform the largest cardiovascular phenotype outcomes study ever.

DETAILED DESCRIPTION:
CONFIRM2 is a retrospective and prospective, open-label, international, multicenter observational registry designed to evaluate associations between CCTA imaging findings and clinical presentation (cross-sectional) and their ability to predict mortality and major adverse cardiac events (longitudinal) in patients with chronic CAD.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Undergoing clinically indicated CCTA with >64-detector row CT
* Signed informed consent, including of release of medical information, long term follow-up and Health Insurance Portability and Accountability Act (HIPAA) documentation

Exclusion Criteria:

* Individuals unable to provide informed consent
* Non-cardiac illness with life expectancy < 2 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable coronary artery disease
Sampling Method: Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Coronary CT Angiography EvaluatioN For Clinical Outcomes | June 2020- June 2022
  Examined the totality of information visualized by coronary CT angiography (CCTA) for optimal refinement of prognostic risk stratification

CONTACTS AND LOCATIONS:
Overall Officials: James K Min, MD, Study Chair — Cleerly, Inc.; Todd Villines, MD, Study Chair — UVA
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feuchtner GM, Lacaita PG, Bax JJ, Rodriguez F, Nakanishi R, Pontone G, Mushtaq S, Buechel RR, Grani C, Patel AR, Singulane CC, Choi AD, Al-Mallah M, Andreini D, Karlsberg RP, Cho G, Rochitte CE, Alasnag M, Hamdan A, Cademartiri F, Maffei E, Marques H, Goncalves Pereira PM, Gupta H, Hadamitzky M, Khalique O, Kalra D, Mills JD, Nurmohamed NS, Knaapen P, Budoff M, Shaikh K, Martin E, German DM, Ferencik M, Oehler AC, Deano R, Nagpal P, Van Assen M, De Cecco CN, Foldyna B, Brendel JM, Cheng VY, Branch K, Bittencourt M, Bhatti S, Polsani V, Wesbey G, Cardoso R, Blankstein R, Delago A, Pursnani A, Alsaid A, Bloom S, Kamperidis V, Barbieri F, Aquino M, Danad I, van Rosendael A. AI-Quantitative CT Coronary Plaque Features Associate With a Higher Relative Risk in Women: CONFIRM2 Registry. Circ Cardiovasc Imaging. 2025 Jun;18(6):e018235. doi: 10.1161/CIRCIMAGING.125.018235. Epub 2025 Mar 31. PMID 40162910